CLINICAL TRIAL: NCT03004170
Title: Telephone Counseling to Enhance the Quality and Safety of Romantic and Sexual Relationships in People Living and Aging With HIV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oregon Health and Science University (Other)
Collaborators: University of Georgia (Other)
Responsible Party: Principal Investigator, Travis Lovejoy, Associate Professor of Psychiatry, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIA-R01AG053081
Record Dates: First submitted 2016-12-20; First posted 2016-12-28 (Estimated); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: HIV Seropositivity
Keywords: HIV; Motivational Interviewing; Telephone; Telehealth; Risky Sex; Unprotected Sex; Condoms; Older Adults
MeSH Terms: conditions — HIV Seropositivity; Unsafe Sex

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome Assessor is blind to participant condition.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tele-Motivational Interviewing Plus Behavioral Skills Training (Experimental): The Telephone-Administered Motivational Interviewing Plus Behavioral Skills Training (teleMI+BST) intervention comprises 5 sessions lasting approximately 45-50 minutes each. Sessions occur in weeks 3, 4, 8, and 12 post-enrollment, with a follow-up booster session in week 24. The Information-Motivation-Behavioral Skills (IMB) Model (Fisher & Fisher, 1992) provides the theoretical framework for behavior change mechanisms of teleMI+BST. The IMB posits that knowledge about condom use practices, condom use motivation, and acquisition and application of requisite condom use skills lead to engagement in condom-protected sex. The focus of this intervention is to help participants process ambivalence about engaging in condomless sex acts that risk HIV transmission.
  Interventions: Behavioral: Telephone-Administered Motivational Interviewing Plus Behavioral Skills Training
- Tele-Coping Effectiveness Training (Active Comparator): The Telephone-Administered Coping Effectiveness Training (teleCET) intervention is the attention-equivalent comparator and also comprises 5 sessions lasting approximately 45-50 minutes each. The teleCET intervention is based on the Lazarus and Folkman Transactional Model of Stress and Coping (Lazarus & Folkman, 1984) and uses cognitive-behavioral principles to: (a) appraise stressor severity, (b) develop problem- and emotion-focused coping skills, (c) determine the match between coping strategies and stressor controllability, and (d) optimize coping through use of social support resources.
  Interventions: Behavioral: Telephone-Administered Coping Effectiveness Training

INTERVENTIONS:
Behavioral: Telephone-Administered Motivational Interviewing Plus Behavioral Skills Training
  Arms: Tele-Motivational Interviewing Plus Behavioral Skills Training
Behavioral: Telephone-Administered Coping Effectiveness Training
  Arms: Tele-Coping Effectiveness Training

SUMMARY:
The purpose of this study is to determine if a brief behavioral intervention delivered over the telephone is effective at reducing occasions of condomless sex in persons living and aging with HIV.

DETAILED DESCRIPTION:
Estimated rates of condomless anal and vaginal intercourse among HIV-positive older adults remain high. Brief motivational interventions delivered face-to-face have demonstrated efficacy at reducing condomless sex in HIV-positive persons. However, these interventions are not contextualized to the unique sexual health needs of HIV-positive older adults. Further, many HIV-positive older adults have difficulty accessing face-to-face services due to transportation, stigma, and other barriers. Telehealth interventions represent one delivery approach that overcomes such barriers.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Have access to a landline or cellular telephone
* Be 50 years of age or older at some point during study participation
* Report engaging in one or more occasions of condomless anal and/or vaginal intercourse with an HIV-negative or unknown HIV serostatus sex partner in the 3 months prior to study enrollment. An exception to this criterion is participants whose HIV viral load is undetectable and whose only condomless sex is in the context of a monogamous sexual relationship with an HIV-negative partner.

Exclusion Criteria:

* Active suicidal ideation as determined by the Patient Health Questionnaire 9-item Depression Module

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in number of condomless sex acts from baseline to 12-month follow-up | Baseline, 12-month follow-up
  Self-reported condomless anal and/or vaginal sex acts with HIV-negative or unknown HIV serostatus sex partners based on the Timeline Followback Interview.

SECONDARY OUTCOMES:
Change in depressive symptom severity from baseline to 12-month follow-up | Baseline, 12-month follow-up
  Self-reported depressive symptom severity using the Patient Health Questionnaire 9-item Depression Module (PHQ-9). This outcome will be assessed among the approximately one-third of participants who report mild levels of depression at study enrollment.

OTHER OUTCOMES:
Change in knowledge of HIV viral load from baseline to 12-month follow-up | Baseline, 12-month follow-up
  Self-reported knowledge of one's HIV viral load status (i.e., test result and date of most recent viral load test)

CONTACTS AND LOCATIONS:
Overall Officials: Travis Lovejoy, PhD, MPH, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
Raw de-identified data will be made publicly available to the scientific community upon request after the trial is complete and data have been published. Data requests should be directed to the study principal investigator.

REFERENCES:
- [Result] Fisher JD, Fisher WA. Changing AIDS-risk behavior. Psychol Bull. 1992 May;111(3):455-74. doi: 10.1037/0033-2909.111.3.455. PMID 1594721
- [Result] Lazarus RS, Susan Folkman. Stress, appraisal, and coping. New York, NY: Springer; 1984.
- [Derived] Kahler J, Heckman TG, Shen Y, Huckans MS, Feldstein Ewing SW, Parsons JT, Phelps A, Sutton M, Holloway J, Lovejoy TI. Randomized controlled trial protocol for project BRIDGE: A telephone-administered motivational interviewing intervention targeting risky sexual behavior in older people living with HIV. Contemp Clin Trials. 2020 Aug;95:106047. doi: 10.1016/j.cct.2020.106047. Epub 2020 May 28. PMID 32474130